CLINICAL TRIAL: NCT03170063
Title: FoxBioNet Pilot Project: SAVE (Synuclein Assay Validation Effort) (SAVE001)
Brief Title: FoxBioNet Pilot Project: SAVE (Synuclein Assay Validation Effort)
Acronym: SAVE001
Status: Completed | Type: Observational
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Collaborators: University Health Network, Toronto (Other); Indiana University (Other); ICON Clinical Research Limited (Unknown)
Responsible Party: Principal Investigator, Connie Marras, Neurologist at Toronto Western Hospital Movement Disorders Centre, University Health Network, Toronto
Other Study IDs: SAVE001
Record Dates: First submitted 2017-05-26; First posted 2017-05-30 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Alpha-Synuclein; Biomarker
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cerebrospinal Fluid, whole blood, serum, and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's Disease Subjects: Up to 30 Parkinson's Disease patients will be enrolled.
  Interventions: Procedure: Procedure/Surgery: Biofluid samplings
- Healthy Controls: Up to 20 healthy controls will be enrolled.
  Interventions: Procedure: Procedure/Surgery: Biofluid samplings

INTERVENTIONS:
Procedure: Procedure/Surgery: Biofluid samplings — Biofluid samplings (blood and cerebrospinal fluid (CSF))

SUMMARY:
The overall objective of this study is to compare the performance of available oligomeric and phosphorylated a-synuclein assay in cerebrospinal fluid and blood.

DETAILED DESCRIPTION:
Specific aims to accomplish this objective are:

1. Assess the reliability of oligomeric and phosphorylated a-synuclein concentration between two different oligomeric and three phosphorylated asynuclein assays.
2. Assess the reliability of the oligomeric and phosphorylated a-synuclein concentrations between laboratories
3. Assess the correlation of oligomeric and phosphorylated a-synuclein concentrations between cerebrospinal fluid and blood.

1.2. Secondary Objectives

1. To assess the ability of the network of pilot sites to efficiently conduct a study involving biosample collection for PD research. Efficiency will be assessed using measures of the time taken to meet specific milestones within the study.
2. To assess the ability of the network to collect high quality biospecimens adhering to agreed-upon protocols.
3. To gauge the willingness of participants to participate in subsequent Fox BioNet studies

ELIGIBILITY:
Inclusion Criteria:

Parkinson's Disease Subjects

* Patients must meet the MDS criteria for Parkinson's disease.
* Disease duration: any
* Male or female age 30 years or older at time of PD diagnosis.

Control Subjects

* Male or female age 30 years or older at Screening.

Exclusion Criteria:

Parkinson's Disease Subjects

* Inability to provide informed consent
* Current treatment with anticoagulants (e.g., coumadin, heparin) that might preclude safe completion of the lumbar puncture.
* Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Participation in a blinded clinical trial of any kind or an unblinded trial of an investigational product that is not currently approved for use in humans.

Control Subjects

* Inability to provide informed consent
* Current treatment with anticoagulants (e.g. coumadin, heparin) that might preclude safe completion of the lumbar puncture.
* Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Participation in a blinded clinical trial of any kind or an unblinded trial of an investigational product that is not currently approved for use in humans.
* The presence of rest tremor, bradykinesia or rigidity.
* The presence of any other neurological sign that in the opinion of the site investigator raises suspicion for an atypical parkinsonian syndrome (e.g. supranuclear gaze palsy)

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 Parkinson's Disease Subjects, and 20 Healthy Controls. Potential participants will be identified by the study sites through their patient population or through Fox Trial Finder.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Oligomeric and PS129 α-syn levels | 3 Months
  CSF, serum, and plasma will be analyzed using oligomeric and pS129 assays. The outcome will be expressed as a concentration of modified (pS129 or oligomeric) synuclein or as a ratio of specific species to total synuclein levels.

SECONDARY OUTCOMES:
Time from IRB submission to approval by central IRB | 3 Months
  To assess time taken from submission of proposal to IRB to approval by the IRB
Time from central IRB approval to site approval (for those sites requiring administrative review) | 3 Months
  To assess time taken from approval by IRB to approval by internal boards for sites.
Time from site selection to contract full execution | 3 Months
  To assess the ability of the network of pilot sites to efficiently conduct a study involving biosample collection for PD research. Efficiency will be assessed using measures of the time taken to meet specific milestones within the study.
Time from site activation to recruitment of 10 participants | 3 Months
  Time taken from site activation to recruitment of 10 participants
Proportion of samples conforming to collection, processing and shipping protocols. | 3 Months
  To assess the ability of the network to collect high quality biospecimens adhering to agreed-upon protocols.
Proportion of participants agreeing to be contacted for future Fox BioNet protocols | 3 Months
  To gauge the willingness of participants to participate in subsequent Fox BioNet studies

CONTACTS AND LOCATIONS:
Overall Officials: Connie Marras, MD, Principal Investigator — University Health Network, Toronto
Locations (5):
- United States (5):
  - Rush University Medical Center, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No